CLINICAL TRIAL: NCT07054411
Title: Hemoglobin Monitoring in Scoliosis Surgery: Comparison of Non-invasive and Invasive Methods
Brief Title: Hemoglobin Monitoring in Scoliosis Surgery
Status: Recruiting | Type: Observational
Sponsor: Erhan Ozyurt (Other Government)
Responsible Party: Sponsor-Investigator, Erhan Ozyurt, Associate Professor, MD, Antalya Training and Research Hospital
Organization: Antalya Training and Research Hospital (Other Government)
Other Study IDs: CEMAL01
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Scoliosis Patients
Keywords: scoliosis; hemoglobin monitoring
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scoliosis patients: Include patients who will undergo elective scoliosis surgery under general anesthesia.
  Interventions: Device: Radical-7 Pulse CO-Oximeter

INTERVENTIONS:
Device: Radical-7 Pulse CO-Oximeter — Rainbow sensors will be placed on the 4th fingertips of the non-dominant hand of the patients and connected to the Radical-7 Pulse CO-Oximeter device and the initial Hb value will be recorded routinely and recorded hourly during the operation. Hemogram samples will be studied in the laboratory. During the operation, every hour and at the end of the operation, SpHb value, Hb, Hct levels in hemogram will be recorded.
  Other Names: Hemogram samples

SUMMARY:
The study is planned to include patients who will undergo elective scoliosis surgery under general anesthesia at the Health Sciences University Antalya Education and Research Hospital. Demographic data including age, gender, height, weight, and ASA score of the patients will be recorded before general anesthesia. ECG, oxygen saturation, and non-invasive blood pressure will be monitored while the patients are lying supine before general anesthesia. An esophageal temperature probe will be placed before being placed in the prone position. All patients will receive standard anesthesia management. After being placed in the prone position, patients will be warmed with heaters containing an air-blowing system during the operation to prevent hypothermia. Anesthesia will be maintained with total intravenous anesthesia as a controlled infusion. Rainbow sensors will be placed on the 4th fingertips of the non-dominant hand of the patients and connected to the Radical-7 Pulse CO-Oximeter device and the initial Hb value will be recorded routinely and recorded hourly during the operation. Hemogram samples will be studied in the laboratory. During the operation, every hour and at the end of the operation, SpHb value, Hb, Hct levels in hemogram will be recorded. At the end of the operation, the amount of intraoperative blood transfusion, the amount of crystalloid and colloid given, the duration of the operation, the duration of anesthesia, urine output, and the need for vasopressors will be routinely recorded. A database will be created in a computer environment from this information.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative hemoglobin ≥ 9 g/dL
* ASA I - III

Exclusion Criteria:

* Patients with hematological disease,
* Uncorrected preoperative anemia (preoperative hemoglobin < 9 g/dL)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who apply to our hospital's orthopedic clinics to undergo elective scoliosis surgery.
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Total Hemoglobin (SpHb) | Before the anesthesia induction
  Total Hemoglobin will be recorded from the monitor
Total Hemoglobin (SpHb) | 1 hour after the anesthesia induction
  Total Hemoglobin will be recorded from the monitor
Total Hemoglobin (SpHb) | 2 hours after the anesthesia induction
  Total Hemoglobin will be recorded from the monitor
Total Hemoglobin (SpHb) | 3 hours after the anesthesia induction
  Total Hemoglobin will be recorded from the monitor
Total Hemoglobin (SpHb) | Through operation completion, an average of 4 hours
  Total Hemoglobin will be recorded from the monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shabaninejad H, Ghadimi N, Sayehmiri K, Hosseinifard H, Azarfarin R, Gorji HA. Comparison of invasive and noninvasive blood hemoglobin measurement in the operating room: a systematic review and meta-analysis. J Anesth. 2019 Jun;33(3):441-453. doi: 10.1007/s00540-019-02629-1. Epub 2019 Mar 20. PMID 30895376